CLINICAL TRIAL: NCT01429246
Title: China Salt Substitute Study in Tibet: Efficacy of Salt Substitute in Reducing Blood Pressure in Hypertensive Adults
Brief Title: China Salt Substitute Study in Tibet
Acronym: CSSS-Tibet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: Peking University (Other); Beijing Jishuitan Hospital (Other); People's Hospital of Dangxiong County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHSN268200900027C
Record Dates: First submitted 2011-08-31; First posted 2011-09-07 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2011-09

CONDITIONS: Hypertension
Keywords: Hypertension; Diet Therapy; Sodium Chloride, Dietary; Tibet; Aged
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Salt (Active Comparator): 100% Sodium Chloride
  Interventions: Dietary Supplement: Regular Salt
- Salt Substitute (Experimental): 65% Sodium Chloride, 25% Potassium Chloride, 10% Magnesium Sulphate)
  Interventions: Dietary Supplement: Salt Substitute

INTERVENTIONS:
Dietary Supplement: Regular Salt — Estimated Household Individual Consumption of 30 grams per day
  Arms: Normal Salt
Dietary Supplement: Salt Substitute — Estimated 30 grams per day per household member
  Arms: Salt Substitute

SUMMARY:
The study was a single-blind randomized controlled trial conducted between February and August 2009 in two townships (Yangbajing and Gongtang) of Dangxiong County, an area at 4300 meters altitude in Tibet. A brief baseline survey and assessment for eligibility was performed before randomization. A total of 282 residents with known hypertension (systolic blood pressure ≥ 140mmHg) were recruited and randomly assigned to intervention or control with stratification by gender and baseline blood pressure. The intervention group received 6-month's supply of salt substitute (68% sodium chloride, 22% potassium chloride and 10% magnesium sulfate heptahydrate) and the control group 6-month's supply of regular salt (100% sodium chloride). After 3-month's intervention, the ones with a blood pressure above 140 mmHg / 90 mmHg will be given low-dose diuretic for further anti-hypertensive therapy. The study hypothesis is that salt-substitute will greatly reduce blood pressure in treated patients when compared to controls. Blood pressure levels were measured at baseline and followed up by trained observers using an automated sphygmomanometer and brief survey on level of compliance, amount of salt consumed, and reasons for non-compliance.

DETAILED DESCRIPTION:
Hypertension is one of the most important risk factors that induce cardiovascular and cerebrovascular disease. Reducing the blood pressure levels of population can not only control the incidence of cardiovascular and cerebrovascular disease effectively, but also reduce the mortality. Anti-hypertension drug therapy has been proven to be an effective method to reduce blood pressure. Dietary sodium restriction and potassium supplementation is the core of dietary approaches to stop hypertension. Tibet is located on the Tibetan Plateau with an average altitude about 4000 meters above sea level. Tibetan diet is rich in meat but poor in vegetables and fruits. Salt intake is quite high due to habitual drinking of salty butter tea. Former national surveys showed a high prevalence of hypertension in Tibet. The investigators conducted this randomized controlled intervention study to test whether the investigators can offer a cost effective way to lower blood pressure and control hypertension in a sample of subjects from Yangbajing and Gongtang in Dangxiong County, Lhasa, Tibet.

A randomized controlled trial was conducted in Yangbajing Township and Gongtang Village in the Dangxiong county , Tibet. A total of 282 hypertensive patients were chosen as study subjects. The regular salt or salt substitution were randomly allocated to the two groups. The whole intervention last for 6 months, with Phase 1 for three months and a following Phase 2 for another three months. For Phase 1, the study subjects were allocated the regular salt or the salt substitute after a randomization. For Phase 2, the study subjects continued the intervention of regular salt or salt substitute while the ones with a blood pressure above 140mmHg/90 mmHg will be given low-dose diuretic for further anti-hypertensive therapy. During the whole intervention period, the study subjects were not informed of what kind of salt they were taking. Blood pressure was the major outcome and would be measured at baseline, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Resident of Yangbajing Township and Gongtang Village in Tibetan Autonomous Region, People's Republic of China
* Mean Systolic Hypertension (≥ 140 mmHg)

Exclusion Criteria:

* Currently taking any potassium supplements (or lives in household where someone does)
* Previously diagnosed kidney disease or gout (or lives in a household where someone does) and physician considered he/she cannot take salt substitute.
* Any person who intended to use salt outside the assigned treatment salt provide in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Mean Systolic Blood Pressure (mmHg) at 6 months | (Baseline compared to 6 months after start of intervention)
  3 Serial in Right Arm with Seated Patients with at least 1 minute between measurements using Omron 751 Automated Cuff.

SECONDARY OUTCOMES:
Percent of patients having blood pressure under control (<140/90 mmHg) | Baseline, and post start of intervention at 3 months and 6 months
Change in Baseline Mean Systolic Blood Pressure (mmHg) at 3 months. | (Baseline compared to 3 months after start of intervention)
  3 Serial in Right Arm with Seated Patients with at least 1 minute between measurements using Omron 751 Automated Cuff

CONTACTS AND LOCATIONS:
Overall Officials: Yangfeng Wu, PhD, Study Director — The George Institute, China (Beijing, CN)
Locations (1):
- Dangxiong People's Hospital, Lhasa, Tibet, China

REFERENCES:
- [Background] Tian HG, Guo ZY, Hu G, Yu SJ, Sun W, Pietinen P, Nissinen A. Changes in sodium intake and blood pressure in a community-based intervention project in China. J Hum Hypertens. 1995 Dec;9(12):959-68. PMID 8746640
- [Background] Hooper L, Bartlett C, Davey SG, Ebrahim S. Advice to reduce dietary salt for prevention of cardiovascular disease. Cochrane Database Syst Rev. 2004;2004(1):CD003656. doi: 10.1002/14651858.CD003656.pub2. PMID 14974027
- [Background] He FJ, MacGregor GA. Effect of longer-term modest salt reduction on blood pressure. Cochrane Database Syst Rev. 2004;(3):CD004937. doi: 10.1002/14651858.CD004937. PMID 15266549
- [Background] China Salt Substitute Study Collaborative Group. Salt substitution: a low-cost strategy for blood pressure control among rural Chinese. A randomized, controlled trial. J Hypertens. 2007 Oct;25(10):2011-8. doi: 10.1097/HJH.0b013e3282b9714b. PMID 17885542
- [Background] Zhou X, Liu JX, Shi R, Yang N, Song DL, Pang W, Li YM. Compound ion salt, a novel low-sodium salt substitute: from animal study to community-based population trial. Am J Hypertens. 2009 Sep;22(9):934-42. doi: 10.1038/ajh.2009.135. Epub 2009 Aug 6. PMID 19661926
- [Background] He FJ, MacGregor GA. Can a low-sodium, high-potassium salt substitute reduce blood pressure in rural Chinese people? Nat Clin Pract Cardiovasc Med. 2008 Apr;5(4):186-7. doi: 10.1038/ncpcardio1122. Epub 2008 Jan 29. No abstract available. PMID 18227813
- [Background] Hu J, Jiang X, Li N, Yu X, Perkovic V, Chen B, Zhao L, Neal B, Wu Y. Effects of salt substitute on pulse wave analysis among individuals at high cardiovascular risk in rural China: a randomized controlled trial. Hypertens Res. 2009 Apr;32(4):282-8. doi: 10.1038/hr.2009.7. Epub 2009 Feb 27. PMID 19262499
- [Background] Li N, Prescott J, Wu Y, Barzi F, Yu X, Zhao L, Neal B; China Salt Substitute Study Collaborative Group. The effects of a reduced-sodium, high-potassium salt substitute on food taste and acceptability in rural northern China. Br J Nutr. 2009 Apr;101(7):1088-93. doi: 10.1017/S0007114508042360. Epub 2008 Aug 19. PMID 18710605
- [Derived] Zhao X, Yin X, Li X, Yan LL, Lam CT, Li S, He F, Xie W, Sang B, Luobu G, Ke L, Wu Y. Using a low-sodium, high-potassium salt substitute to reduce blood pressure among Tibetans with high blood pressure: a patient-blinded randomized controlled trial. PLoS One. 2014 Oct 22;9(10):e110131. doi: 10.1371/journal.pone.0110131. eCollection 2014. PMID 25338053